CLINICAL TRIAL: NCT06551506
Title: A Prospective, Randomized, Open-label Phase 4 Study of the Immunology and Safety of Maternal RSV Vaccination (ABRYSVO (TM)), Infant Nirsevimab (BEYFORTUS (TM)) Immunization, or Both Products During the First Year of Life
Brief Title: The Immunology and Safety of Maternal RSV Vaccination (ABRYSVO), Infant Nirsevimab (BEYFORTUS) Immunization, or Both Products
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0003; 5UM1AI148684-04 (NIH)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-02-11

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: ABRYSVO; BEYFORTUS; Immunology; Infants; Nirsevimab; Respiratory syncytial virus; RSV; RSVpreF
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — abrysvo; nirsevimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1A (Experimental): Mother receives 120 mcg/0.5ml of maternal RSVpreF (ABRYSVO) administered intramuscularly once during 32 0/7 to 36 6/7 weeks GA and infant does NOT receive nirsevimab. N= 50.
  Interventions: Biological: Abrysvo
- Group 1B (Experimental): Mother receives 120 mcg/0.5ml of maternal RSVpreF (ABRYSVO) administered intramuscularly once during 32 0/7 to 36 6/7 weeks GA and infant receives one dose of nirsevimab (BEYFORTUS) 50mg/0.5mL if body weight <5kg or 100mg/mL if body weight is >= 5kg at birth. N= 50.
  Interventions: Biological: Abrysvo; Biological: Beyfortus
- Group 1C (Experimental): Mother receives 120 mcg/0.5ml of maternal RSVpreF (ABRYSVO) administered intramuscularly once during 32 0/7 to 36 6/7 weeks GA and infant receives one dose of nirsevimab (BEYFORTUS) 50mg/0.5mL if body weight <5kg or 100mg/mL if body weight is >= 5kg at 3-month . N= 50.
  Interventions: Biological: Abrysvo; Biological: Beyfortus
- Group 2 (Experimental): Mother does NOT receive maternal RSVpreF and infant receives one dose of nirsevimab (BEYFORTUS) 50mg/0.5mL if body weight <5kg or 100mg/mL if body weight is >= 5kg at birth . N= 50.
  Interventions: Biological: Beyfortus

INTERVENTIONS:
Biological: Abrysvo — A maternal RSV vaccine based on the prefusion F protein administered during pregnancy
  Arms: Group 1A; Group 1B; Group 1C
Biological: Beyfortus — A passive, long-acting monoclonal antibody to Respiratory syncytial virus (RSV) administered to infants
  Arms: Group 1B; Group 1C; Group 2

SUMMARY:
Respiratory Syncytial Virus (RSV) is the leading cause of lower respiratory tract infections (LRTIs) in infants and young children. It is also a leading cause of mortality in children <5 years of age worldwide. Until recently, no Food and Drug Administration (FDA)-approved vaccines were available to prevent RSV infection. The only prophylactic product for RSV prevention recommended for infants was the monoclonal antibody palivizumab, but administration was limited to those with extreme prematurity, chronic lung disease, or hemodynamically significant congenital heart disease. However, in 2023, the FDA approved two products designed to prevent RSV lower respiratory tract disease (LRTD) in all infants: an active RSV vaccine based on the prefusion F protein (RSVpreF, ABRYSVO, Pfizer) administered during pregnancy, and a passive, long-acting monoclonal antibody (nirsevimab-alip [henceforth referred to as nirsevimab], BEYFORTUS, AstraZeneca) administered to infants at birth or at the start of their first RSV season. Both products were evaluated in Phase 3 pivotal clinical trials and have high efficacy in preventing LRTD caused by RSV in infants. Although there is no established correlate of protection against RSV, antibodies have been associated with protection across multiple studies. The clinical development plan for the products did not include comprehensive evaluations of the magnitude and durability of the immune response, nor were the two products tested in a single trial. This study is a prospective, randomized, open-label Phase 4 study with the primary objective of evaluating the magnitude and durability of RSV-specific neutralizing antibodies in infants through 12 months of life following either maternal RSV vaccination, infant nirsevimab administration, or both products combined.

DETAILED DESCRIPTION:
Respiratory Syncytial Virus (RSV) is the leading cause of lower respiratory tract infections (LRTIs) in infants and young children. It is also a leading cause of mortality in children <5 years of age worldwide. Until recently, no Food and Drug Administration (FDA)-approved vaccines were available to prevent RSV infection in infants. Only the monoclonal antibody palivizumab was available to high-risk infants, but administration was limited to those with extreme prematurity, chronic lung disease, or hemodynamically significant congenital heart disease. However, in 2023, the FDA approved two products designed to prevent RSV lower respiratory tract disease (LRTD) in all infants: an active RSV vaccine based on the prefusion F protein (RSVpreF, ABRYSVO, Pfizer) administered during pregnancy and a passive, long-acting monoclonal antibody (nirsevimab, BEYFORTUS, AstraZeneca) administered to infants at birth or at the start of the first RSV season. Both products were evaluated in Phase 3 pivotal clinical trials and were found to have high efficacy in the prevention of RSV LRTD in infants. However, the magnitude and durability of antibody responses following administration of the products have not been directly compared. This is important because although there are no well-established correlates of protection against RSV, serum antibodies have been associated with protection across multiple studies.

Furthermore, the added benefit of administering both products to an infant has not been characterized. While cost-effectiveness analyses have demonstrated that administration of both products to the same mother-infant dyad is not cost-effective or indicated, it is likely that some infants may receive both products inadvertently, and still others may benefit from both. These include infants born to women who may not have mounted an adequate antibody response to vaccination (e.g., due to immunocompromise, prematurity, or insufficient time from vaccination to delivery) or who may have had impaired antibody transfer across the placenta (e.g., due to placental pathology). It also includes high-risk infants (e.g., with prematurity or chronic lung disease) who may benefit from an interval dose of nirsevimab for protection in the setting of waning antibodies and off-season RSV circulation. Thus, understanding the safety and immunology of administration of both products vs. either product alone is of clinical and public health importance. These knowledge gaps underlie the objectives for this study.

Primary objective: To evaluate the magnitude and durability of RSV-specific neutralizing antibodies in infants through 12 months of life following either maternal RSV vaccination, infant nirsevimab administration, or both products combined. Secondary objective: 1) To describe the safety among infants exposed to maternal RSV vaccination alone, infant nirsevimab administration alone, or both products combined. 2) To describe the tolerability among infants following administration of nirsevimab. 3)To describe the transplacental transfer of RSV-specific antibodies from mother to infant among individuals who received RSV vaccination during pregnancy and those who did not. 4) To describe the magnitude and durability of RSV-specific antibodies in maternal milk through 12 months of life among individuals who received RSV vaccination during pregnancy and those who did not. 5) To describe the magnitude and durability of RSV-specific antibodies through 12 months post-delivery in mothers among the study groups. 6) To evaluate the magnitude and durability of RSV-specific binding antibodies in infants through 12 months of life among the study groups.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years of age at time of enrollment with an uncomplicated singleton pregnancy who are at no known increased risk for complications per clinical judgement of the investigator
2. Understands and agrees to comply with all study procedures
3. Willing and able to provide consent for study participation for themselves and their infant prior to initiation of any study procedures
4. In good health, as determined by the medical history and clinical judgment of the investigator Note: Healthy volunteers with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.
5. Intention to deliver at a hospital or birthing facility where study procedures can be performed
6. Eligible to receive either product per the FDA package inserts. (Maternal RSVpreF from 32 0/7 to 36 6/7 weeks gestational age (GA) from September 1 to March 31)

Exclusion Criteria:

1. Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the study
2. Any condition which, in the opinion of the investigators, may pose a health risk for the participant or interfere with the evaluation of study objectives
3. Maternal bleeding diathesis, or any condition which may contraindicate intramuscular injection
4. Maternal known or suspected congenital or acquired disease that impairs the immune system, including functional asplenia or immunosuppression due to underlying illness or treatment
5. Maternal receipt of immunosuppressive drugs or biologic agents within 30 days prior to enrollment (This includes oral or parenteral corticosteroids. The use of inhaled/nebulized, intra-articular, intrabursal, or topical (skin, eye, ears) steroids are permitted. This does not include RhoGAM)
6. Maternal conditions known to impair transplacental transfer of maternal antibodies (e.g., placental pathology, hypergammaglobulinemia, HIV)
7. Maternal history of GBS or other potentially immune-mediated medical condition (PIMMC)
8. Maternal history of severe adverse reaction or anaphylaxis to ABRYSVO or its components
9. Maternal history of preterm birth (<34 weeks GA)
10. Current pregnancy complicated by uncontrolled hypertension, pre-eclampsia, or eclampsia
11. Previous receipt of ABRYSVO or other approved or investigational RSV vaccine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of serum RSV A and B neutralizing antibodies in infants | Through Day 366
  GMT of RSV A and B neutralizing antibodies in infant serum at Day 1, 43, 91, 181, and 366. Day 1 infant specimen represents infant cord blood or serum (if unable to collect cord blood). Mother-infant pairs will be randomized 1:1 to either Day 43 or Day 91 blood collection.

SECONDARY OUTCOMES:
Frequency and relatedness of serious adverse events (SAEs) in each study arm (infants only) | Through Day 181
  Number of participants that experienced SAEs by relatedness in each study arm
Frequency and severity of unsolicited Grade 3 or higher related adverse events (AEs) | Through 30 days following each nirsevimab dose
  Number of participants that experienced unsolicited Grade 3 or higher related AEs by severity
Frequency and severity of medically attended adverse events (MAAEs) | Through 30 days following each nirsevimab dose
  Number of participants that experienced MAAEs by severity
Geometric mean titer (GMT) of RSV A and B neutralizing antibodies in cord blood | Day 1
  GMT of RSV A and B neutralizing antibodies in cord blood
Geometric mean titer (GMT) of RSV pre-F binding IgG antibodies in cord blood | Day 1
  GMT of RSV pre-F binding IgG antibodies in cord blood
Geometric mean titer (GMT) of RSV pre-F binding IgG antibodies in mothers | Through Day 366
Geometric mean titer (GMT) of serum RSV A and B neutralizing antibodies | Through Day 366
Geometric mean titer (GMT) of serum RSV A and B neutralizing antibodies in mothers | Day 1
  GMT of serum RSV A and B neutralizing antibodies in mothers that had infant cord blood collected
Geometric mean titer (GMT) of serum RSV pre-F binding IgG antibodies in infants | Through Day 366
  GMT of RSV pre-F binding IgG antibodies in infant serum. Day 1 infant specimen represents infant cord blood or serum (if unable to collect cord blood). Mother-infant pairs will be randomized 1:1 to either Day 43 or Day 91 blood collection.
Geometric mean titer (GMT) of serum RSV pre-F binding IgG antibodies in mothers | Day 1
  GMT of serum RSV pre-F binding IgG antibodies in mothers that had infant cord blood collected
Occurrence of local solicited adverse reactions | Through 7 days following each nirsevimab dose
  Number of participants that experienced any local solicited adverse reactions including injection site erythema/redness, injection site edema/induration, and injection site pain/tenderness
Occurrence of systemic solicited adverse reactions | Through 7 days following each nirsevimab dose
  Number of participants that experienced any systemic solicited adverse reactions including fever (axillary), sleepiness/fatigue, irritability/crying, and loss of appetite

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - New York University School of Medicine - Langone Medical Center - Vaccine Center, New York, New York
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio
  - University of Pittsburgh - Medicine - Infectious Diseases, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT06551506/ICF_000.pdf